CLINICAL TRIAL: NCT03606486
Title: Lavage of the Uterine Cavity for Diagnosis of Ovarian Carcinomas
Brief Title: Lavage of the Uterine Cavity for Diagnosis of Ovarian Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: University of Washington (Other)
Collaborators: Minnesota Ovarian Cancer Alliance (Other)
Responsible Party: Principal Investigator, Barbara Norquist, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10019; NCI-2018-01242 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1001786 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: High Grade Ovarian Serous Adenocarcinoma; Stage III Ovarian Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Therapeutic Irrigation; Papanicolaou Test; Vaginal Smears

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (pap smear, uterine lavage, tumor sample) (Experimental): Participants undergo pap smear, uterine lavage, and collection of tumor sample during a planned surgery. DNA is then extracted from the samples and sequenced for TP53 mutations using Crispr-Duplex sequencing.
  Interventions: Other: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Device: Lavage; Other: Pap Smear

INTERVENTIONS:
Other: Biospecimen Collection — Undergo collection of tumor sample and blood draw
Other: Laboratory Biomarker Analysis — Correlative studies
Device: Lavage — Undergo uterine lavage
  Other Names: Irrigation
Other: Pap Smear — Undergo pap smear
  Other Names: Cervical Smear Preparation; Cervical Smear Procedure; Pap Smear Procedure; Pap Test; Papanicolaou Smear Procedure; Papanicolaou Test; Vaginal Smears

SUMMARY:
The goal of this project is to develop a minimally invasive test to detect ovarian cancer, by searching for mutations from the tumor in samples obtained from the cervix (Pap smears), and from the uterus (uterine lavage) in participants with advanced ovarian cancer and in participants with increased risk of ovarian cancer due to inherited mutations, such as BRCA or BRCA2 (among others).

Pap smear and uterine lavage samples will be collected while the participant is under anesthesia for planned debulking surgery. A novel, highly sensitive and accurate technique, Crispr-Duplex sequencing, will be used to detect tumor associated mutations in TP53 (the most commonly mutated gene in ovarian cancer) within these samples. These results will be compared to sequencing results in the tumor itself for comparison, and Pap and uterine lavage will be compared to each other to determine the optimal test. Ultimately, the goal is to use the results of this study to plan a larger study including women without cancer who are at either increased risk or normal risk of ovarian cancer, for use in early detection.

DETAILED DESCRIPTION:
OUTLINE:

Participants undergo pap smear, uterine lavage, and collection of tumor sample during a planned surgery. DNA is then extracted from the samples and sequenced for TP53 mutations using Crispr-Duplex sequencing.

ELIGIBILITY:
Inclusion Criteria:

* With suspected advanced ovarian cancer or genetic predisposition to malignant neoplasm of the ovary
* Planned surgery
* Have a uterus and no history of tubal occlusion

Exclusion Criteria:

* Unable to speak English
* Unable to provide informed consent
* Prior hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara S. Norquist, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Rosana Risques, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (Pap Smear, Uterine Lavage, Tumor Sample): Participants undergo pap smear, uterine lavage, and collection of tumor sample during a planned surgery. DNA is then extracted from the samples and sequenced for TP53 mutations using Duplex sequencing.
  Biospecimen Collection: Undergo collection of tumor sample
  Laboratory Biomarker Analysis: Correlative studies
  Lavage: Undergo uterine lavage
  Pap Smear: Undergo pap smear
Period: Overall Study
Arm/Group | Diagnostic (Pap Smear, Uterine Lavage, Tumor Sample)
Started | 52
Completed | 47
Not Completed | 5
Not completed — Unable to collect sample | 5

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Pap Smear, Uterine Lavage, Tumor Sample)
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants] — >=18 years
  Participants
    <=18 years | 0
    Between 18 and 65 years | 34
    >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 45
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: 20 Ovarian Cancer Participants With Detection of Associated TP53 Mutation in Uterine Lavage
Description: In participants with ovarian cancer, we compared the detection of TP53 mutations in the uterine lavage specimen compared to the ovarian cancer.
Time Frame: A single point in time after sample collection, no follow-up of participants is done
Population: We were able to enroll 20 participants who ended up having ovarian cancer. We recruited less than expected due to the COVID19 pandemic and increased use of neoadjuvant chemotherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Pap Smear, Uterine Lavage, Tumor Sample)
Number analyzed (Participants) | 20
Participants | 13

ADVERSE EVENTS:
Time Frame: At the time of sample collection (during surgery).
Arm/Group | Diagnostic (Pap Smear, Uterine Lavage, Tumor Sample)
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03606486/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT03606486/SAP_001.pdf